CLINICAL TRIAL: NCT00885963
Title: A Phase II Study of Oral Sapacitabine in Patients With Previously Treated Non-Small Cell Lung Cancer
Brief Title: A Study of Oral Sapacitabine in Patients With Previously Treated Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Limitation in financial resources.
Sponsor: Cyclacel Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYC682-08
Record Dates: First submitted 2009-03-31; First posted 2009-04-22 (Estimated); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sapacitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sapacitabine (Experimental): Part A (lead-in phase): Two dosing schedules, i.e., once daily (q.d.) or twice daily (b.i.d.) x 5 days/week x 2 weeks every 3 weeks will be evaluated.
  Part B (Phase 2): Receive the recommended phase 2 dose of once daily or twice daily dosing schedule derived from Part A.
  Interventions: Drug: sapacitabine

INTERVENTIONS:
Drug: sapacitabine — twice daily by mouth for 7 days or once daily by mouth for 5 days/week x 2 weeks every 21 days
  Other Names: CYC682

SUMMARY:
A phase II study to evaluate the safety and efficacy of oral sapacitabine in previously treated advanced non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is an open label, single arm, phase II study to evaluate the safety and efficacy of oral sapacitabine administered twice daily for 5 consecutive days every week for 2 weeks followed by 7-day rest in patients who have had one prior chemotherapy regimen for advanced Non-Small Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent NSCLC
* Age of 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Measurable disease according to RECIST
* Had only 1 prior chemotherapy regimen for metastatic or recurrent disease; patients who have received more than one prior chemotherapy regimens may participate in Part A of the study only.
* Adequate bone marrow function
* Adequate renal function
* Adequate liver function
* At least 3 weeks from prior systemic treatments including investigational anti-cancer therapy; at least 7 days from prior radiation therapy; and have recovered from prior toxicities
* At least 3 weeks from major surgery
* Patient must be able to swallow capsules
* Agree to practice effective contraception during the entire study period and for one month after being discontinued from the study unless documentation of infertility exists. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and willingness to sign the informed consent form

Exclusion Criteria:

* NSCLC histology contains a component of small cell lung cancer
* Previously untreated CNS metastasis or progressive CNS metastasis documented by MRI scan performed at 4 weeks or longer after the last treatment for CNS metastasis
* Currently receiving radiotherapy, biological therapy, or any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Cancer other than NSCLC that has been treated with chemotherapy or biological therapy in the past 5 years with the exception of adequately treated in situ cervical cancer, and basal or squamous cell skin cancer; patients who received only hormonal therapy in the neoadjuvant or adjuvant setting in the past 5 years may participate in this study
* Pregnant or lactating women
* Known to be HIV-positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-12-01 (Actual); Primary Completion 2013-08-13 (Actual); Study Completion 2013-12-23 (Actual)

PRIMARY OUTCOMES:
the rate of response and stable disease | after cycle 2, 4, 7 and every 3 cycles thereafter
  complete response or partial response and stable disease

SECONDARY OUTCOMES:
progression-free survival | 1.5 years
  Time until disease progression
duration of response | 1.5 years
  Observed response time
duration of stable disease | 1.5 years
  Observed time of the disease state within -30% and +10% of the baseline
overall survival | 1.5 years
  Median survival time of the overall patient population in the study

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bonomi, M.D., Study Chair — Rush University Medical Center
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania